CLINICAL TRIAL: NCT00562601
Title: Apheresis Procedures to Obtain Plasma or Leukocytes for In Vitro Studies
Brief Title: LCI Apheresis to Obtain Plasma or White Blood Cells
Status: Terminated | Type: Observational
Why Stopped: Closed by the Sponsor/DSMB/IRB
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 870163; 87-I-0163
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Apheresis
Keywords: Leukapheresis; Plasmapheresis; Lymphocytes; Neutrophils

SUMMARY:
This study will collect blood plasma and white blood cells from individuals using a procedure called apheresis. Apheresis is a method of collecting larger quantities of certain blood components than can safely be collected through a simple blood draw or blood donation process. The blood components will be used in laboratory research studies to investigate aspects of infectious and immunologic allergic diseases.

Patients 7 years of age and older who are currently enrolled in a NIH clinical research protocol may participate in this study. (Children between the ages of 2 and 6 may participate if they will benefit clinically from undergoing apheresis.) Family members of patients and normal healthy volunteers will also be enrolled.

* For all adults and children weighing 55 pounds or more. Blood is drawn through a needle placed in an arm vein and circulated through a cell separator machine. The plasma and white cells are extracted, and the red cells are returned to the donor through a needle in the other arm. The procedure takes from 1 to 2 hours.
* For children weighing less than 55 pounds. One unit (1 pint) of blood is drawn through a needle placed in an arm vein, similar to donating a pint of whole blood. The red blood cells are separated from the rest of the blood and returned to the donor through the same needle. This procedure requires only one needlestick and takes about 30 to 45 minutes to complete. In some circumstances, the procedure must be repeated one or more times in order to obtain large enough quantities of plasma or cells for study.

DETAILED DESCRIPTION:
In order to carry out in vitro research procedures on the plasma or leukocyte components of blood, it is often necessary to obtain larger quantities of plasma or leukocytes than can be safely obtained by simple phlebotomy. These components can be easily and safely obtained using apheresis procedures performed in the Apheresis Clinic of the Department of Transfusion Medicine, Clinical Center. This protocol is specifically designed to conform to the requirements of the Apheresis Clinic for donors to have apheresis procedures, but the protocol in itself is not a research protocol. Patients must first be admitted to another approved clinical research protocol of the NIAID before they may have the apheresis procedures described in this protocol. Family members and healthy volunteers may undergo apheresis using only this protocol, without the necessity for entry into any other protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to undergo apheresis procedures, patients will be admitted to active clinical research protocols approved by the ICRS. Relatives and normal volunteers may undergo apheresis without first being on an active clinical protocol. Women who are pregnant and normal children will not be studied.

In order to undergo apheresis procedures, as a minimum, patients, family members and control subjects must have a recent history and physical examination, as well as CBC and differential count. Appropriate chemistry and coagulation studies will be performed when clinically indicated. If indicated, a pregnancy test may be performed.

Patients and volunteers undergoing apheresis will be tested against HIV, HBsAg and HCV, if not tested in the previous year.

To be eligible for apheresis for research purposes, children must be at least 7 years old, weigh 25 kilograms, have adequate peripheral access to insert needles for apheresis, and be able to undergo apheresis without sedation. If children between the ages of seven and twelve years are to undergo apheresis, a third party not otherwise involved with the protocol ; e.g., Bioethicist, Patient Advocate, must talk with the child independently to ensure that the child understands the procedure and freely agrees to participate. This protocol alone is not intended for general study of patients, but only as an adjunct protocol to allow for apheresis procedures.

For patients, the following minimal criteria are required to undergo the procedure:

* Adequate peripheral venous access;
* No need for sedation;
* Weight greater than 25 kg;
* Hematocrit greater than 27%;
* Platelet count greater than 75,000/microL;
* For patients, the hematological values have to be current (up to a week before the procedure).

Healthy volunteers and relatives will have a CBC performed up to 4 weeks before the procedure. In order to be able to undergo the procedure, they must fulfill all of the below:

* Hemoglobin greater than 11 g/dL for males and greater than 10 g/dL for females;
* Platelet count greater than 150,000 microL;
* WBC greater than 3.5 x 10(3) /microL;
* MCV above 80;
* Negative HIV, HCV and HBsAg serologies in the past year.

EXCLUSION CRITERIA:

Patients will not undergo apheresis procedures if they have cardiovascular instability, severe anemia, inadequate venous access, severe coagulation disorder, are pregnant, or have any other condition which the attending physician or Apheresis Clinic staff considers a contraindication to the procedure.

For children, exclusion criteria include age less than 7 years, weigh less than 25 kilograms, inadequate peripheral access to insert needles for apheresis, and unable to undergo apheresis without sedation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 1988-03-28 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bolan CD, Yau YY, Cullis HC, Horwitz ME, Mackall CL, Barrett AJ, Malech HL, Rehak NN, Wayne AS, Leitman SF. Pediatric large-volume leukapheresis: a single institution experience with heparin versus citrate-based anticoagulant regimens. Transfusion. 2004 Feb;44(2):229-38. doi: 10.1111/j.1537-2995.2004.00668.x. PMID 14962314
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1987-I-0163.html